CLINICAL TRIAL: NCT02831777
Title: CareTaker Self-Calibration Validation
Acronym: Self_Cal
Status: Completed | Type: Observational
Sponsor: CareTaker Medical LLC (Industry)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: SELF_CAL_001
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Blood Pressure
Keywords: non-invasive blood pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: non-invasive blood pressure monitor — Equivalence of CareTaker blood pressure to classical sphygmomanometry

SUMMARY:
The goal of the study is to test the capability of the CareTaker monitor to calibrate its continuous blood pressure readings independently. Currently the device requires another approved blood pressure monitor to provide a starting calibration.

The new control module enables the CareTaker to perform a pressure sweep of the internal pressure in the finger cuff. The resulting data is analyzed using a combination of pulse analysis/oscillometry approach.

DETAILED DESCRIPTION:
The specific objective of this project was to demonstrate the CareTaker's ability to perform self-calibration to the same performance standard as its predicate device. That device demonstrated efficacy by showing substantial equivalence to the performance of classical sphygmomanometry using a Riva-Rocci/Korotkoff (RRK) measurement on the brachial artery, meeting a bias of at least 5 mmHg and a standard deviation of 8 mmHg across 3 paired readings from at least 85 patients, for a total of at least 255 paired readings.

The study was performed at the University of Virginia Medical Center in Charlottesville, Virginia. UVA's Institutional Review Board approved (#18686) and supervised the study for subjects who were University of Virginia hospital patients and staff > 18 years of age and who were able to give verbal consent.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age, who are able and willing to participate and have given verbal assent

Exclusion Criteria:

* Unable to give verbal assent
* <18 years of age
* No or poor finger pulse, as determined through visual inspection for ischemic hands

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be UVA patients/staff, > 18 years of age, who are able and willing to participate and have given verbal assent
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Performance comparison | 8 minutes for 3 paired readings
  Comparison with performance of classical sphygmomanometry using a Riva-Rocci/Korotkov (RRK) measurement on the brachial artery, meeting a bias of at least 5 mmHg and a standard deviation of 8 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Baruch, PhD, Principal Investigator — CareTaker Medical LLC

IPD SHARING:
Plan to Share IPD: Undecided